CLINICAL TRIAL: NCT00697736
Title: Cardiac Repercussion of Systemic Sclerodermias : Detection of Infra-clinical Abnormalities by Analysis of the Myocardic Regional Function Using Myocardial Tissular Doppler Mode.
Brief Title: Cardiac Repercussion of Systemic Sclerodermias
Acronym: HTAP-SCLERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2005.392
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2015-11

CONDITIONS: Systemic Scleroderma
Keywords: Systemic Scleroderma; Echocardiography
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Echocardiography with myocardial tissular Doppler mode — Echocardiography with myocardial tissular Doppler mode during rest and exercise on a table equipped with a cyclo-ergometer

SUMMARY:
Systemic sclerodermia is a connectivity characterized by multiple visceral impairments, in particular pulmonary, which can lead to the development of a Pulmonary Arterial Hypertension (PAHT).

In one hand, this PAHT is an evolutionary turn in symptomatology and prognosis, and on the other hand, the tracking and the analysis of its effects on the right ventricular function are difficult with the conventional techniques.

So, the analysis of the right ventricular function appears capital, because:

* it is recognized like an essential determinant of the symptoms and effort capacity,
* its prevalence, physiopathology and prognostic values remain unknown in this pathology,
* its interest in the starting of the treatment remains to be specified.

The aim of this trial is to identify in a population of 150 patients presenting a systemic scleroderma without PAHT:

* the incidence of a right ventricular dysfonction, evaluated by the analysis of the myocardic regional function with myocardial tissular Doppler mode,
* the physiopathology of this damage by correlation with the tests of respiratory function and the not invasive hemodynamic datas at rest and exercise.
* the prognosis value of the abnormalities of the right ventricular function by a follow-up of these patients over a 5 years period.

This trial should allowed to define the place of the new right ventricular function markers in the evaluation of the functional consequences, the forecast and perhaps the care of systemic sclerodermic patients.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 years and 75 years

* Having a maximum speed of IT < 2.8 m/sec.
* Having read and understood the information note and having signed the informed consent form.
* And :

  * Either carrying a systemic sclerodermia satisfying the criteria of American College of Rheumatology (the presence of a major criteria or two minor criterias is required for the systemic diagnosis of sclerodermia):

    * Major criteria: proximal sclerodermia defined by a bilateral cutaneous sclerosis extending beyond the metacarpophalangeal and metatarsophalangeal joint.
    * Minor criteria: pulpar sclerodactylia, pulpar canker or scars, pulmonary fibrosis on thoracic radiography.
  * Or presenting CREST syndrome, with at least 4 of the 5 following criterias :

    * subcutaneous calcinosis,
    * syndrome of Raynaud,
    * attack oesophagienne,
    * sclerodactylia,
    * telangiectasis.

Exclusion Criteria:

* Over 75 years
* Having a maximum speed of TI > 2.8 m/sec.
* Patient affected by a connectivitis other than a sclerodermia : mixed connectivity, disseminated erythematous lupus, inflammatory idiopathic myopathy, rheumatoïd polyarthritis.
* Patient carrying a sclerodermia complicated by:
* renal failure (clearance > 30 ml - Cockraft)
* recent heart failure (< 2 months)
* cardiac valvular attack, dilated, hypertrophic or restrictive cardiomyopathy, constrictive pericarditis, chronic pulmonary heart or antecedent of myocarditis
* Coronaropathy objectified by stenosis or simple coronary irregularities on the coronarography or antecedent of myocardial infarction
* Chronic respiratory handicap with another origin than sclerodermia
* Unsigned informed consent form
* Patient with mental or psychiatric disorders, unable or unwilling to comply with protocol requirements.
* Patient treated with intraveinous derived of prostacyclin within 1 month before inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2007-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To measure the incidence of right ventricular dysfonction evaluated by analysis of the regional myocardic function with myocardial tissular Doppler mode | each year for 5 years

SECONDARY OUTCOMES:
To define the potential place of new regional myocardic function markers in the evaluation of the cardiac repercussion of systemic scleroderma and to correlate these markers with clinical, functional and hemodynamic parameters. | each year for five years
To detect an eventual prognostic role of regional myocardic function parameters which could allow to an earlier screening of the patients being able to receive a pulmonary vasodilator treatment before the rest PAHT occurrence . | each year for five years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

REFERENCES:
- [Result] Thuny F, Lovric D, Schnell F, Bergerot C, Ernande L, Cottin V, Derumeaux G, Croisille P. Quantification of myocardial extracellular volume fraction with cardiac MR imaging for early detection of left ventricle involvement in systemic sclerosis. Radiology. 2014 May;271(2):373-80. doi: 10.1148/radiol.13131280. Epub 2014 Jan 15. PMID 24475856